CLINICAL TRIAL: NCT04766060
Title: Indocyanine Green Enhanced Fluorescent Angiography: Can it Predict Anastomotic Leakage (AL) After Recto-sigmoid Resection for Malignancy, and Are we Able to Evaluate the Findings? -A Small Multi-centre Trial Study
Brief Title: Indocyanine Green Fluorescent Imaging in Robotic Assisted Rectosigmoidal Resection; a Multicenter Assessment of Interobserver Variation and Comparison With Computer-based Pixel Analysis
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Pernille Larsen, Medical Doctor, Odense University Hospital
Other Study IDs: PLarsen
Record Dates: First submitted 2021-02-18; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Colorectal Cancer; Anastomotic Leak
MeSH Terms: conditions — Colorectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Fluorescent Imaging — Fluorescense imaging used to evaluate blood perfusion

SUMMARY:
A serious complication to colorectal surgery is anastomotic leakage (AL). AL increases post-operative mortality, decreases long-term survival, reduces the functional result and reduces qual-ity of life. Studies suggest that performing an indocyanine-green enhanced fluorescent angi-ography (ICGeFA), blood perfusion in the bowel can be visualised. It is suggested that using this procedure the relative risk of AL is reduced about 54-67%.

With this project we wish to evaluate the feasibility of the procedure, and, if proven feasible, to plan further studies evaluating the procedure.

DETAILED DESCRIPTION:
Colorectal cancer is one of the most common cancer-diagnosis in Denmark. In 2014, 5186 pa-tients with colorectal cancer were registered. 1674 patients had cancer in the rectum and 1316 in the sigmoid colon. 668 patients underwent surgery with low anterior resection (LAR) and primary anastomosis, and 850 patients had a sigmoid resection with primary anastomosis.

A serious complication is anastomotic leakage (AL). In 2014 a total of 67 (10%) patients were registered with AL.

In general AL increases the post-operative mortality, decreases long-term survival and reduces the functional result and thereby reduces quality of life.

Due to the possible severity of AL all measures possible should be taken to ensure an early diag-nosis and timely treatment, as this has been shown to reduce morbidity and mortality. The symp-toms of AL are uncharacteristic; the diagnosis cannot only rely on the development of clinical symptoms. However, specific clinical scoring symptoms, measuring C-reactive protein (CRP) and radiologic examinations are proven useful.

Treatment of AL varies with the degree of leakage, from conservative treatment with rectal lavage, endo-VAC therapy, drainage of abscesses, re-laparoscopy or laparotomy with a diverting stoma, and finally to break down the anastomosis and creating a temporary or permanent colostomy, all procedures with or without antibiotic treatment.

It is essential that surgeons continuously strive to improve the operative technique with regard to anastomosis construction. Many factors influence the anastomotic healing: instrumentation error, tension on the anastomosis, bacterial contamination, etc. An important factor to ensure most opti-mal conditions in anastomotic healing is to ensure sufficient blood-supply/oxygen tension.

The surgeon evaluate so-called surrogates of bowel perfusion (evaluation of colour, mesenteric pulsation and arterial bleeding) prior to form the anastomosis, but studies have demonstrated that surgeon's intraoperative judgment in predicting of anastomotic leakage AL has an extremely low sensitivity and specificity.

Studies suggest that performing an indocyanine-green enhanced fluorescent angiography (ICGeFA), the blood perfusion in the bowel can be visualised. It is suggested that by evaluating perfusion of bowel ends, and, if needed, doing a re-resection, the risk of anastomotic leakage can be diminished. It is suggested that evaluating the anastomosis with ICG-FA and revising the anas-tomosis if necessary, the relative risk reduction of AL is about 54-67%. Several studies in robotic and laparoscopic colorectal surgery, confirms feasibility of using ICGeFA, also showing promising results in evaluating the bowel perfusion. Most studies and a newly published systematic review conclude that there is great need for larger controlled studies or randomised trails.

The primary objective with this study is to evaluate the feasibility of using ICGeFA in colorectal surgery and to evaluate if the surgeon's interpretation is dose and time dependent. Secondary ob-jective is to establish a nationwide research team, joining all the Robotic Surgery Centres in Den-mark for future research.

Last we wish to identify the optimal design for a further study, evaluating whether ICG is a helpful tool in diminishing the risk of anastomotic leakage.

ELIGIBILITY:
Inclusion Criteria:

* robotic surgery for rectal cancer and cancers located low in the sigmoid bowel

Exclusion Criteria:

* Allergy of iodide
* Pregnancy
* Lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, older than 18, undergoing robotic surgery for rectal cancer and cancers located low in the sigmoid bowel, <25 cm form the anal verge.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with anastomotic leakage and evaluation of fluorescent imaging in these patients | 30 days
  Primary surgeons peroperative evaluation of fluoresence

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Fyn, Denmark

REFERENCES:
- [Derived] Larsen PO, Nerup N, Andersen J, Dohrn N, Klein MF, Brisling S, Salomon S, Andersen PV, Moller S, Svendsen MBS, Rahr HB, Iversen LH, Gogenur I, Qvist N, Ellebaek MB. Anastomotic perfusion assessment with indocyanine green in robot-assisted low-anterior resection, a multicenter study of interobserver variation. Surg Endosc. 2023 May;37(5):3602-3609. doi: 10.1007/s00464-022-09819-1. Epub 2023 Jan 9. PMID 36624218